CLINICAL TRIAL: NCT00244725
Title: A Dose Ranging Trial for the Evaluation of the Safety, Tolerability and Efficacy of Odiparcil in the Prevention of Venous Thromboembolism Following Total Knee Replacement Surgery
Brief Title: Odiparcil For The Prevention Of Venous Thromboembolism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: ITI101711
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-03

CONDITIONS: Deep Vein Thrombosis; Fibrillation, Atrial; Venous Thromboembolism; Pulmonary Embolism
Keywords: deep vein thrombosis; total knee replacement; PE; Venous thromboembolism; DVT; pulmonary embolism; VTE
MeSH Terms: conditions — Venous Thrombosis; Atrial Fibrillation; Venous Thromboembolism; Pulmonary Embolism | interventions — odiparcil; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Odiparcil
Drug: Warfarin
Drug: Coumadin
  Other Names: Odiparcil; Warfarin

SUMMARY:
Odiparcil is being studied to determine if it can prevent blood clots from forming after a total knee replacement and also to prove that odiparcil is safe.

ELIGIBILITY:
Inclusion Criteria:

* Women must be unable to have children.
* Will have a total knee replacement.

Exclusion Criteria:

* Allergic to any X-ray dye.
* Allergies or reactions to warfarin or coumadin.
* Previous VTE (venous thromboembolism) or deep vein thrombosis (DVT).
* On anticoagulation therapy.
* Renal impairment.
* Participated in any clinical trial in the past 30 days.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 961 (Actual)
Dates: Start 2005-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (91):
- United States (40):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Banning, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Yuba City, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Lonetree, Colorado
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Sarsota, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Warren, Michigan
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Altoona, Pennsylvania
  - GSK Investigational Site, Camp Hill, Pennsylvania
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Lubbock, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Huntington, West Virginia
  - GSK Investigational Site, Marshfield, Wisconsin
- Australia (7):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Southport, Queensland
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Geelong, Victoria
  - GSK Investigational Site, Ringwood East, Victoria
  - GSK Investigational Site, Windsor, Victoria
- GSK Investigational Site, Porto Alegre, Rio Grande do Sul, Brazil
- Canada (12):
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Ajax, Ontario
  - GSK Investigational Site, Don Mills, Ontario
  - GSK Investigational Site, Newmarket, Ontario
  - GSK Investigational Site, North York, Ontario
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Scarborough Village, Ontario
  - GSK Investigational Site, Waterloo, Ontario
  - GSK Investigational Site, Charlottetown, Prince Edward Island
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sainte Jerome, Quebec
- India (2):
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Secunderabad
- Israel (4):
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Tel Aviv
- GSK Investigational Site, Riga, Latvia
- Lithuania (3):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Klaipėda
  - GSK Investigational Site, Vilnius
- Poland (4):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Sosnowiec
  - GSK Investigational Site, Wroclaw
- Russia (5):
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Kurgan
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Mosocow
  - GSK Investigational Site, Rostov-on-Don
- South Africa (3):
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Centurion
  - GSK Investigational Site, Pretoria
- Ukraine (4):
  - GSK Investigational Site, Cherkasy
  - GSK Investigational Site, Dnipro
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Vinnitsa
- United Kingdom (5):
  - GSK Investigational Site, Birmingham, West Midlands
  - GSK Investigational Site, Bournmouth
  - GSK Investigational Site, Fife
  - GSK Investigational Site, London
  - GSK Investigational Site, Wigan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male or female participants >=35 years of age with scheduled for primary elective unilateral total knee arthroplasty were recruited at 82 centers from 13 countries. The study was conducted between 28 September 2005 and 27 September 2006.
Pre-assignment Details: A total of 958 participants were randomized into the study. Two participants each from the treatment arm Odiparcil 250 milligram (mg), and Odiparcil 375 mg did not receive the study medication. Therefore, the intent to treat (ITT) population was comprised of 954 participants.
Groups:
- Odiparcil MR 250 mg Tablet: Eligible participants received Odiparcil modified release (MR) 250 mg tablet at every 12 hours interval (Q12h)for the duration of 10 ± 2 days of double-blind treatment period.
- Odiparcil MR 375 mg Tablet: Eligible participants received Odiparcil MR 375 mg tablet at Q12h for the duration of 10 ± 2 days of double-blind treatment period.
- Odiparcil MR 500 mg Tablet: Eligible participants received Odiparcil MR 500 mg tablet at Q12h for the duration of 10 ± 2 days of double-blind treatment period.
- Warfarin INR 2.0 to 3.0: Eligible participants received overencapsulated warfarin 1 mg and 5 mg as guided by investigator to adjust warfarin to a target International Normalized Ratio (INR) of 2.0 to 3.0 according to the investigators practice or participant status for the duration of 10 ± 2 days of double-blind treatment period.
Period: Overall Study
Arm/Group | Odiparcil MR 250 mg Tablet | Odiparcil MR 375 mg Tablet | Odiparcil MR 500 mg Tablet | Warfarin INR 2.0 to 3.0
Started | 237 | 245 | 239 | 237
Completed | 214 | 226 | 215 | 216
Not Completed | 23 | 19 | 24 | 21
Not completed — Lost to Follow-up | 3 | 4 | 9 | 2
Not completed — Withdrawal by Subject | 9 | 7 | 7 | 8
Not completed — Not meet treatment eligibility criteria | 1 | 2 | 0 | 0
Not completed — Physician Decision | 3 | 0 | 1 | 2
Not completed — Adverse Events | 3 | 1 | 4 | 4
Not completed — Withdrwal by participant | 1 | 0 | 0 | 1
Not completed — Liver function test abnormality | 2 | 0 | 0 | 1
Not completed — Sponsor withdrew the participant | 1 | 0 | 0 | 1
Not completed — Mediciation Error | 0 | 1 | 0 | 0
Not completed — Rehab Refused to allow participantion | 0 | 1 | 0 | 0
Not completed — Headache | 0 | 1 | 0 | 0
Not completed — Received prohibited medication | 0 | 1 | 0 | 1
Not completed — Confirmed venous thromboembolism (VTE) | 0 | 1 | 0 | 0
Not completed — Administrative reason | 0 | 0 | 1 | 0
Not completed — Vomit | 0 | 0 | 1 | 0
Not completed — Failed to follow-up | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Odiparcil MR 250 mg Tablet: Eligible participants received Odiparcil MR 250 mg tablet, Q12h for the duration of 10 ± 2 days of double-blind treatment period.
- Odiparcil MR 375 mg Tablet: Eligible participants received Odiparcil MR 375 mg tablet, Q12h for the duration of 10 ± 2 days of double-blind treatment period.
- Odiparcil MR 500 mg Tablet: Eligible participants received Odiparcil MR 500 mg tablet, Q12h for the duration of 10 ± 2 days of double-blind treatment period.
- Warfarin INR 2.0 to 3.0: Eligible participants received overencapsulated warfarin 1 mg and 5 mg as guided by investigator to adjust warfarin to a target INR of 2.0 to 3.0 according to the investigators practice or participant status for the duration of 10 ± 2 days of double-blind treatment period.
- Total: Total of all reporting groups
Arm/Group | Odiparcil MR 250 mg Tablet | Odiparcil MR 375 mg Tablet | Odiparcil MR 500 mg Tablet | Warfarin INR 2.0 to 3.0 | Total
Number analyzed (Participants) | 235 | 243 | 239 | 237 | 954
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.1 (9.53) | 65.3 (8.93) | 64.5 (8.68) | 66.1 (9.30) | 65.5 (9.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 156 | 155 | 150 | 611
  Male | 85 | 87 | 84 | 87 | 343
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 18 | 17 | 20 | 12 | 67
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian - Central/South Asian Heritage | 3 | 1 | 3 | 3 | 10
  Asian - East Asian Heritage | 0 | 1 | 1 | 0 | 2
  Asian - South East Asian Heritage | 0 | 0 | 0 | 1 | 1
  White - Arabic/North African Heritage | 1 | 0 | 1 | 0 | 2
  White - White/Caucasian/European Heritage | 212 | 224 | 210 | 220 | 866
  Mixed Race | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Total VTE Event Over 10 ± 2 Days of Treatment
Description: Participants were assessed for VTE at all study visits and at the end of study (Day 10±2) or at early withdrawal. Any participant who remained asymptomatic for VTE at the end of the study did not receive a mandatory bilateral venogram following at least 8 days on study medication. Participants who were withdrawn early and had been objectively confirmed to have a VTE event by a method other than venography were not required to undergo venography. A participant was included in the Independent Central Adjudication Committee (ICAC)-adjudicated incidence of total VTE if he/ she experienced any of adjudicated asymptomatic deep vein thrombosis (DVT) at early withdrawal or after 8-12 days of study treatment and no later than 1 day after end of study treatment, adjudicated symptomatic DVT or pulmonary embolism (PE) at any time during study treatment or death adjudicated to be related to VTE during study treatment.
Time Frame: Up to Visit 7 (10 ± 2 days of treatment)
Population: ITT population comprised of all participants who were randomized and received at least one dose of study treatment. Total number of participants with objectively confirmed symptomatic VTE, venographically detected VTE at early withdrawal or an evaluable venogram at study completion were used for analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Odiparcil MR 250 mg Tablet | Odiparcil MR 375 mg Tablet | Odiparcil MR 500 mg Tablet | Warfarin INR 2.0 to 3.0
Number analyzed (Participants) | 164 | 169 | 160 | 157
Percentage of participants | 45.1 [37.4 to 53.1] | 44.4 [36.8 to 52.2] | 41.3 [33.5 to 49.3] | 31.2 [24.1 to 39.1]
Statistical Analysis 1: Comparison: Odiparcil MR 250 mg Tablet vs Warfarin INR 2.0 to 3.0; Test type: Superiority or Other; p = 0.012, Fisher Exact; Risk Ratio (RR) = 1.45, 95% CI 2-sided [1.1 to 1.9]
Statistical Analysis 2: Comparison: Odiparcil MR 375 mg Tablet vs Warfarin INR 2.0 to 3.0; Test type: Superiority or Other; p = 0.017, Fisher Exact; Risk Ratio (RR) = 1.42, 95% CI 2-sided [1.1 to 1.9]
Statistical Analysis 3: Comparison: Odiparcil MR 250 mg Tablet vs Warfarin INR 2.0 to 3.0; Test type: Superiority or Other; p = 0.080, Fisher Exact; Risk Ratio (RR) = 1.32, 95% CI 2-sided [1.0 to 1.8]

2. Secondary Outcome: Percentage of Participants With Proximal DVT Over 10 ± 2 Days of Treatment
Description: Proximal DVT is defined as DVT in or above the popliteal vein. A participant was considered to have had an asymptomatic evaluable venogram if the ICAC answer to the DVT question was 'Yes' or 'No', and to have had an adjudicated asymptomatic DVT if the answer was 'Yes'. A participant who reported symptoms of DVT was considered to had an adjudicated objectively confirmed symptomatic DVT if the ICAC answer to the question 'Was a symptomatic DVT identified?' was 'Yes' and the event happened no more than 12 days after start of study treatment (unless exemption for extended treatment was granted by the medical monitor) and no more than 1 day after end of study treatment. In both asymptomatic and symptomatic DVT, the participant was considered to had a proximal DVT if either of the ICAC answers to the questions 'Left proximal' and 'Right proximal' was 'DVT'. Percentage of participants with proximal DVT over 10 ± 2 days of treatment were reported.
Time Frame: Up to 12 days
Population: ITT population. The participants from ITT population who were with objectively confirmed symptomatic VTE, venographically detected VTE at early withdrawal or an evaluable venogram at completion of study treatment were used for the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Odiparcil MR 250 mg Tablet | Odiparcil MR 375 mg Tablet | Odiparcil MR 500 mg Tablet | Warfarin INR 2.0 to 3.0
Number analyzed (Participants) | 164 | 169 | 160 | 157
Percentage of participants
  Asymptomatic, Proximal DVT | 1.8 [0.4 to 5.3] | 1.8 [0.4 to 5.1] | 4.4 [1.8 to 8.8] | 0.6 [0.0 to 3.5]
  Symptomatic, Proximal DVT | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.2] | 0.6 [0.0 to 3.4] | 0.0 [0.0 to 2.3]
  Total, Proximal DVT | 1.8 [0.4 to 5.3] | 1.8 [0.4 to 5.1] | 5.0 [2.2 to 9.6] | 0.6 [0.0 to 3.5]

3. Secondary Outcome: Percentage of Participants With Distal DVT Over 10 ± 2 Days of Treatment
Description: A participant was considered to have had an asymptomatic evaluable venogram if the ICAC answer to the DVT question was 'Yes' or 'No', and to have had an adjudicated asymptomatic DVT if the answer was 'Yes'. A participant who reported symptoms of DVT was considered to had an adjudicated objectively confirmed symptomatic DVT if the ICAC answer to the question 'Was a symptomatic DVT identified?' was 'Yes' and the event happened no more than 12 days after start of study treatment (unless exemption for extended treatment was granted by the medical monitor) and no more than 1 day after end of study treatment. In both asymptomatic and symptomatic DVT, the participant was considered to had a distal DVT if either of the investigator's answers to the questions 'Left distal' and 'Right distal' is 'DVT'.
Time Frame: Up to 12 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of paticipants
Arm/Group | Odiparcil MR 250 mg Tablet | Odiparcil MR 375 mg Tablet | Odiparcil MR 500 mg Tablet | Warfarin INR 2.0 to 3.0
Number analyzed (Participants) | 164 | 169 | 160 | 157
Percentage of paticipants
  Asymptomatic, Distal DVT | 42.1 [34.4 to 50.0] | 43.8 [36.2 to 51.6] | 38.8 [31.2 to 46.8] | 30.6 [23.5 to 38.4]
  Symptomatic, Distal DVT | 1.8 [0.4 to 5.3] | 0.0 [0.0 to 2.2] | 0.6 [0.0 to 3.4] | 0.0 [0.0 to 2.3]
  Total, Distal DVT | 43.9 [36.2 to 51.9] | 43.8 [36.2 to 51.6] | 39.4 [31.8 to 47.4] | 30.6 [23.5 to 38.4]

4. Secondary Outcome: Percentage of Participants With PE Over 10 ± 2 Days of Treatment
Description: Participant who reported symptoms of PE were considered to have had an adjudicated objectively confirmed symptomatic PE if the ICAC answer to the question 'Was a PE identified?' was 'Yes'. E was characterized as fatal PE non-fatal PE and total PE events. Data has been presented for fatal PE non-fatal PE and total PE events over 12 days.
Time Frame: Up to 12 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Odiparcil MR 250 mg Tablet | Odiparcil MR 375 mg Tablet | Odiparcil MR 500 mg Tablet | Warfarin INR 2.0 to 3.0
Number analyzed (Participants) | 164 | 169 | 160 | 157
Percentage of participants
  Fatal PE | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3] | 0.0 [0.0 to 2.3]
  Non-fatal PE | 1.2 [0.1 to 4.3] | 0.6 [0.0 to 3.3] | 0.0 [0.0 to 2.3] | 0.6 [0.0 to 3.5]
  Total PE | 1.2 [0.1 to 4.3] | 0.6 [0.0 to 3.3] | 0.0 [0.0 to 2.3] | 0.6 [0.0 to 3.5]

5. Secondary Outcome: Number of Death Due to VTE Over 10 ± 2 Days of Treatment
Description: A participant was considered dead from an adjudicated VTE-related cause if the death classification was recorded as 'Fatal PE'. A participant was considered to have died from an investigator-assessed VTE-related cause if the investigator's death classification was recorded as 'Fatal PE'. Number of death due to VTE over 10 ± 2 days of treatment were reported.
Time Frame: Up to 12 days
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Odiparcil MR 250 mg Tablet | Odiparcil MR 375 mg Tablet | Odiparcil MR 500 mg Tablet | Warfarin INR 2.0 to 3.0
Number analyzed (Participants) | 164 | 169 | 160 | 157
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With Total Asymptomatic VTE Over 10 ± 2 Days of Treatment
Description: A participant was included in the Independent Central Adjudication Committee (ICAC)-adjudicated incidence of total VTE if experienced any of adjudicated asymptomatic deep vein thrombosis (DVT) at early withdrawal or after 8-12 days of study treatment and no later than 1 day after end of study treatment, adjudicated symptomatic DVT or PE at any time during study treatment or death adjudicated to be related to VTE during study treatment. A participant was considered to have had an asymptomatic evaluable venogram if the ICAC answer to the DVT question was 'Yes' or 'No', and to have had an adjudicated asymptomatic DVT if the answer was 'Yes'. The participant was considered to had a proximal DVT if either of the investigator's answers to the questions 'Left distal' and 'Right distal' is 'DVT'. The participant was considered to had a distal DVT if either of the investigator's answers to the questions 'Left distal' and 'Right distal' is 'DVT'.
Time Frame: Up to 12 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Odiparcil MR 250 mg Tablet | Odiparcil MR 375 mg Tablet | Odiparcil MR 500 mg Tablet | Warfarin INR 2.0 to 3.0
Number analyzed (Participants) | 164 | 169 | 160 | 157
Percentage of participants | 42.1 [34.4 to 50.0] | 43.8 [36.2 to 51.6] | 40.0 [32.3 to 48.0] | 30.6 [23.5 to 38.4]

7. Secondary Outcome: Percentage of Total Symptomatic VTE Over 10 ± 2 Days of Treatment
Description: A participant who reported symptoms of DVT was considered to had an adjudicated objectively confirmed symptomatic DVT if the ICAC answer to the question 'Was a symptomatic DVT identified?' was 'Yes' and the event happened no more than 12 days after start of study treatment (unless exemption for extended treatment was granted by the medical monitor) and no more than 1 day after end of study treatment. The participant was considered to had a proximal DVT if either of the investigator's answers to the questions 'Left distal' and 'Right distal' was 'DVT'. The participant was considered to had a distal DVT if either of the investigator's answers to the questions 'Left distal' and 'Right distal' was 'DVT'. Percentage of participants with total symptomatic (distal and proximal) VTE over 10 ± 2 days of treatment were reported.
Time Frame: Up to 12 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Perentage of participants
Arm/Group | Odiparcil MR 250 mg Tablet | Odiparcil MR 375 mg Tablet | Odiparcil MR 500 mg Tablet | Warfarin INR 2.0 to 3.0
Number analyzed (Participants) | 164 | 169 | 160 | 157
Perentage of participants | 1.8 [0.4 to 5.3] | 0.0 [0.0 to 2.2] | 1.3 [0.2 to 4.4] | 0.0 [0.0 to 2.3]

8. Secondary Outcome: Concentration of Trough Anti-IIa Activity Over the Duration of Treatment and Follow-up
Description: In all participants, additional 3 milliliter of blood was collected at the time of other blood sampling as follow: Baseline, Day 3 (predose, 2, 4, 8, 10, and 12 hours post dose), Day 5 (predose), and Day 10 (predose) or early withdrawal from study medication for the assessment of anti-factor IIa activity. Samples were collected in 3.8% sodium citrate tubes and immediately chilled in ice. Plasma were centrifuged and frozen at approximately -20ºC until time of shipment to the regional central laboratory. Concentration of Trough Anti-IIa Activity over the duration of treatment and follow-up were reported.
Time Frame: Up to 68 days
Population: ITT population.
Measure: Geometric Mean (Standard Deviation); unit: Microgram per millilitre (mcg/ml)
Arm/Group | Odiparcil MR 250 mg Tablet | Odiparcil MR 375 mg Tablet | Odiparcil MR 500 mg Tablet | Warfarin INR 2.0 to 3.0
Number analyzed (Participants) | 235 | 243 | 239 | 237
Microgram per millilitre (mcg/ml)
  Day 3, n= 224, 221, 223, 220 | 2.44 (1.944) | 3.15 (2.667) | 3.75 (2.702) | 0.26 (0.041)
  Day 5, n= 201, 207, 215, 203 | 1.73 (1.456) | 2.43 (1.924) | 3.07 (2.440) | 0.27 (0.099)
  Day 10, n= 179, 197, 199, 181 | 1.45 (1.298) | 2.23 (1.830) | 2.45 (2.042) | 0.25 (0.020)
  Early Withdraw On-therapy, n= 13, 8, 10, 17 | 1.73 (1.286) | 3.73 (2.684) | 2.49 (3.072) | 0.29 (0.159)
  14 Day FU, n= 16, 11, 5, 9 | 0.95 (1.086) | 1.16 (1.431) | 1.02 (1.652) | 0.30 (0.109)
  Early Withdraw 14 Day FU, n= 13, 15, 6, 13 | 0.46 (0.376) | 0.74 (0.767) | 0.60 (0.666) | 0.25 (0.008)
  28 Day FU, n= 0, 1, 0, 1 | NA (NA) — Participants were not analyzed at this time point. | 0.25 (NA) — Standard deviation was not derived as only one participant was available at the time of analysis analyzed. | NA (NA) — Participants were not analyzed at this time point. | 0.25 (NA) — Standard deviation was not derived as only one participant was available at the time of analysis analyzed.
  Early Withdraw 28 Day FU, n=0, 1, 0, 1 | NA (NA) — Participants were not analyzed at this time point. | 0.25 (NA) — Standard deviation was not derived as only one participant was available at the time of analysis analyzed. | NA (NA) — Participants were not analyzed at this time point. | 0.25 (NA) — Standard deviation was not derived as only one participant was available at the time of analysis analyzed.

9. Secondary Outcome: Percentage of Participants With Major Bleeds Over 10 ± 2 Days of Treatment
Description: A participant was included in the ICAC-adjudicated incidence of major bleeding if participant experienced an adjudicated major bleed up to 12 days after the start of study treatment and no later than 1 day after end of study treatment. Major bleed was defined as clinically overt bleeding, 1) Clinical overt bleeding: clinically apparent bleeding or signs and/or symptoms suggestive of bleeding with confirmatory imaging studies (e.g., ultrasound, computed tomography) 2. Critical Site Involvement: Intracranial, retroperitoneal, intra-ocular, intraspinal, pericardial. 3. Decrease in Hgb > 2 g/dL from baseline, 4. Transfusion of > 2 units of packed RBCs, 5. Medical or Surgical Intervention for the Reported Bleed, 6. Fatal Bleed. If the event satisfied one of the above criteria.
Time Frame: Up to 12 days
Population: ITT Population. The participants from ITT population who completed study treatment (Day-10 visit) or reported a major bleed by the time of early withdrawal were used for the analysis
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Odiparcil MR 250 mg Tablet | Odiparcil MR 375 mg Tablet | Odiparcil MR 500 mg Tablet | Warfarin INR 2.0 to 3.0
Number analyzed (Participants) | 205 | 217 | 222 | 203
Percentage of participants | 0.0 [0.0 to 1.8] | 0.0 [0.0 to 1.7] | 0.9 [0.1 to 3.2] | 1.0 [0.1 to 3.5]

10. Secondary Outcome: Percentage of Participants With VTE and/or Major Bleeding Over 10±2 Days of Treatment
Description: A participant was included in the ICAC-adjudicated incidence of major bleeding if experienced an adjudicated major bleed up to 12 days after the start of study treatment and no later than 1 day after end of study treatment. Percentage of participants with VTE and/or major bleeding over 10±2 days of treatment were reported.
Time Frame: Up to 12 days
Population: ITT population. The participants from ITT population who were efficacy evaluable or reported a major bleed or VTE by the time of early withdrawal were used for the analysis
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Odiparcil MR 250 mg Tablet | Odiparcil MR 375 mg Tablet | Odiparcil MR 500 mg Tablet | Warfarin INR 2.0 to 3.0
Number analyzed (Participants) | 164 | 169 | 160 | 157
Percentage of participants
  VTE and/or major bleed | 45.1 [37.4 to 53.1] | 44.4 [36.8 to 52.2] | 42.5 [34.7 to 50.6] | 32.5 [25.2 to 40.4]
  VTE and major bleed | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3] | 0.0 [0.0 to 2.3]
  VTE with no major bleed | 45.1 [37.4 to 53.1] | 44.4 [36.8 to 52.2] | 41.3 [33.5 to 49.3] | 31.2 [24.1 to 39.1]
  Major bleed with no VTE | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.2] | 1.3 [0.2 to 4.4] | 1.3 [0.2 to 4.5]
  No VTE and no major bleed | 54.9 [46.9 to 62.6] | 55.6 [47.8 to 63.2] | 58.1 [50.1 to 65.9] | 68.2 [60.3 to 75.4]

11. Secondary Outcome: Percentage of Participants With Total VTE Any Time After Start of Treatment
Description: Participants were assessed for VTE at all study visits and at the end of the study (Day 10±2) or at early withdrawal. Any participant who remained asymptomatic for VTE at the end of the study were received a mandatory bilateral venogram. Participants who were withdrawn early and had been objectively confirmed to have a VTE event by a method other than venography were not required to undergo venography. A participant was included in the ICAC-adjudicated incidence of total VTE if experienced any of adjudicated asymptomatic DVT at early withdrawal or after 8-12 days of study treatment and no later than 1 day after end of study treatment, adjudicated symptomatic DVT or PE at any time during study treatment or death adjudicated to be related to VTE during study treatment. Percentage of participants with total VTE any time after start of treatment were reported.
Time Frame: Up to Visit 9 (Day 28 post treatment)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percenatge of participants
Arm/Group | Odiparcil MR 250 mg Tablet | Odiparcil MR 375 mg Tablet | Odiparcil MR 500 mg Tablet | Warfarin INR 2.0 to 3.0
Number analyzed (Participants) | 170 | 179 | 171 | 168
Percenatge of participants | 46.5 [38.8 to 54.3] | 45.8 [38.4 to 53.4] | 43.3 [35.7 to 51.1] | 30.4 [23.5 to 37.9]

12. Secondary Outcome: Percentage of Participants With Elevated Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Direct Bilirubin (DB) and Total Bilirubin (TB) by 2 Fold and 3 Fold From Upper Normal Limits (ULN) Any Time On-treatment
Description: The ranges (low concern value; high concern value) for AST (none; > 3 fold upper normal limit (ULN) ), ALT (none; >3 fold ULN), total bilirubin (none; >= 34.2 micromole per litre [umol/L]), Direct bilirubin (none; >= 34.2 umol/L). Percentage of participants with elevated values by 2 fold and 3 fold from ULN any time on-treatment were reported.
Time Frame: Up to 12 days
Population: ITT population. Number of participants were available at the time of analysis were included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Odiparcil MR 250 mg Tablet | Odiparcil MR 375 mg Tablet | Odiparcil MR 500 mg Tablet | Warfarin INR 2.0 to 3.0
Number analyzed (Participants) | 231 | 235 | 236 | 234
Percentage of participants
  ALT, >=2xULN | 4.8 [2.4 to 8.4] | 3.8 [1.8 to 7.1] | 3.8 [1.8 to 7.1] | 5.6 [3.0 to 9.3]
  ALT, >=3xULN | 0.9 [0.1 to 3.1] | 2.6 [0.9 to 5.5] | 0.4 [0.0 to 2.3] | 2.1 [0.7 to 4.9]
  AST, >=2xULN | 2.6 [1.0 to 5.6] | 3.4 [1.5 to 6.6] | 3.8 [1.8 to 7.1] | 4.7 [2.4 to 8.3]
  AST, >=3xULN | 0.0 [0.0 to 1.6] | 0.9 [0.1 to 3.1] | 0.4 [0.0 to 2.3] | 1.7 [0.5 to 4.3]
  Total Billirubin, >=2xULN | 0.0 [0.0 to 1.6] | 0.4 [0.0 to 2.3] | 0.4 [0.0 to 2.3] | 0.0 [0.0 to 1.6]
  Total Billirubin, >=3xULN | 0.0 [0.0 to 1.6] | 0.0 [0.0 to 1.6] | 0.0 [0.0 to 1.6] | 0.0 [0.0 to 1.6]
  Direct Billirubin, >=2xULN | 0.4 [0.0 to 2.4] | 0.4 [0.0 to 2.3] | 0.4 [0.0 to 2.3] | 0.9 [0.1 to 3.1]
  Direct Billirubin, >=3xULN | 0.4 [0.0 to 2.4] | 0.4 [0.0 to 2.3] | 0.0 [0.0 to 1.6] | 0.0 [0.0 to 1.6]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAE) and non-serious adverse events (nSAEs) were collected up to follow-up visit (Visit 9, Day 28±2 days after study medication discontinuation). On-treatment nSAEs were reported.
Description: ITT population was used for analysis.
Arm/Group | ODIPARCIL MR 250 mg Tablet | ODIPARCIL MR 375 MG TABLET | ODIPARCIL MR 500 MG TABLET | WARFARIN INR 2.0 TO 3.0
Serious Adverse Events (participants affected / at risk) | 14/235 | 11/243 | 16/239 | 9/237
Other Adverse Events (participants affected / at risk) | 124/235 | 120/243 | 122/239 | 104/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ODIPARCIL MR 250 mg Tablet (N=235) | ODIPARCIL MR 375 MG TABLET (N=243) | ODIPARCIL MR 500 MG TABLET (N=239) | WARFARIN INR 2.0 TO 3.0 (N=237)
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 1 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis acute (Infections and infestations) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Bleeding time abnormal (Investigations) | 1 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0 | 0 — General disorders and administration site conditions
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 — General disorders and administration site conditions
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ODIPARCIL MR 250 mg Tablet (N=235) | ODIPARCIL MR 375 MG TABLET (N=243) | ODIPARCIL MR 500 MG TABLET (N=239) | WARFARIN INR 2.0 TO 3.0 (N=237)
Nausea (Gastrointestinal disorders) | 27 (28) | 35 (36) | 40 (41) | 33 (36)
Pyrexia (General disorders) | 40 (42) | 28 (30) | 29 (29) | 34 (34)
Constipation (Gastrointestinal disorders) | 29 (30) | 25 (25) | 26 (26) | 29 (31)
Oedema peripheral (General disorders) | 27 (30) | 23 (27) | 28 (36) | 25 (35)
Anaemia postoperative (Injury, poisoning and procedural complications) | 20 (20) | 21 (21) | 24 (24) | 19 (19)
Vomiting (Gastrointestinal disorders) | 19 (19) | 15 (15) | 21 (21) | 13 (14)
Body temperature increased (Investigations) | 18 (20) | 21 (21) | 13 (13) | 13 (13)
Insomnia (Psychiatric disorders) | 17 (18) | 11 (11) | 16 (17) | 13 (13)
Tachycardia (Cardiac disorders) | 11 (12) | 12 (12) | 19 (19) | 12 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (11) | 14 (14) | 10 (10) | 9 (9)
Dizziness (Nervous system disorders) | 8 (8) | 9 (9) | 14 (16) | 11 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (9) | 10 (10) | 13 (14) | 9 (11)
Contusion (Injury, poisoning and procedural complications) | 7 (8) | 13 (14) | 8 (10) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.